CLINICAL TRIAL: NCT07327619
Title: A Multicenter, Randomized, Double-blind, Active-Controlled, Parallel, Phase Ⅲ Study to Evaluate the Efficacy and Safety of Meropenem and Pralurbactam for Injection Compared to Ceftazidime and Avibactam Sodium for Injection in Subjects With Hospital-acquired and Ventilator-associated Bacterial Pneumonia
Brief Title: A Study to Evaluate the Efficacy and Safety of Meropenem and Pralurbactam in HABP/VABP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FL058-303
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Hospital-acquired Bacterial Pneumonia and Ventilator-associated Bacterial Pneumonia
MeSH Terms: interventions — Meropenem; avibactam, ceftazidime drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem and Pralurbactam (Experimental)
  Interventions: Drug: Meropenem and Pralurbactam
- Ceftazidime-avibactam (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam

INTERVENTIONS:
Drug: Meropenem and Pralurbactam — 3g，q8h，120min infusion
  Arms: Meropenem and Pralurbactam
Drug: Ceftazidime-avibactam — 2.5g，q8h，120min infusion
  Arms: Ceftazidime-avibactam

SUMMARY:
This study is to evaluate the efficacy and safety of Meropenem and Pralurbactam for Injection in Subjects with HABP/VABP. The primary objective is to demonstrate non-inferiority of Meropenem and Pralurbactam to Ceftazidime and Avibactam Sodium for Injection. This study is a randomized, double-blind, active-controlled study. The total duration of the study will be approximately 32 days including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female participants ≥18 and ≤80 years of age

  2. have a diagnosis of HAP/VAP.

  3. have systemic signs and respiratory signs or symptoms of HAP/VAP.

  4. New or worsening infiltrate on chest X-ray/CT obtained within 48 hours prior to screening.

  5. The estimated survival time is at lest 28 days.

Exclusion Criteria:

* 1. Diagnosed or suspected CAP, Atypical pneumonias, Viral pneumonia or Chemical pneumonia.

  2. The total duration of antibiotic exposure for antibiotics whose administration begins in the 72 hours is longer than 24 hours.

  3. Acute Physiology and Chronic Health Evaluation (APACHE) II score >30.

  4. Allergic to any carbapenem, cephalosporin, penicillin, metronidazole disodium phosphate, other beta-lactam drugs or other beta-lactamase inhibitors and their auxiliary materials.

  5. Those who have a history of drug abuse or drug abuse within 6 months before screening.

  6. Those who participated in other clinical trials within 28 days before randomization and used any test drugs or medical devices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Died Due to Any Cause Description: Due to Day 14，Proportion of Participants Who Died Due to Any Cause in mITT | Day 14